CLINICAL TRIAL: NCT00606008
Title: A Phase II Trial of Sutent (Sunitinib; SU011248) for Recurrent Anaplastic Astrocytoma and Glioblastoma Multiforme
Brief Title: A Phase II Trial of Sutent (Sunitinib; SU011248) for Recurrent Anaplastic Astrocytoma and Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14916
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-09

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma
Keywords: Sutent
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sutent Treatment (Experimental): Sutent was administered daily for 4 weeks at a dose of 50 mg followed by a 2 week study drug free break.
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — Initially, patients were started on sunitinib at a dose of 50 mg daily. If 50 mg daily resulted in unacceptable toxicity, 2 dose modifications were allowed (to 37.5 and to 25 mg daily, if necessary). Study patients who could not tolerate 25 mg daily of sunitinib were taken off study.
  Other Names: Sutent; SU011248

SUMMARY:
We are asked patients to take part in this study because they had recurrent (returned) (1st or 2nd) anaplastic astrocytoma (AA) or glioblastoma multiforme (GBM).

The purposes of this study are:

* To see if Sutent has any change on the patient and their cancer.
* To see if Sutent will slow or stop the growth of their tumor.
* To measure the safety of Sutent. Sutent is Food and Drug Administration (FDA) approved to treat patients with a gastrointestinal stromal tumor after the disease worsened while taking another medicine called imatinib mesylate or when imatinib mesylate cannot be taken. Sutent is also FDA approved to treat patients with advanced renal cell carcinoma. At this time, it is not known whether Sutent will improve symptoms, or help patients with this disease live longer.

DETAILED DESCRIPTION:
Trial patients received sunitinib 50 mg daily for 4 weeks without regard to meals, followed by a 2-week rest period. This 6-week regimen constituted 1 cycle. Patients were treated for up to 9 cycles [~ year) or until disease progression or death or if persistent toxicities occurred. Complete blood count with differential, complete metabolic profile, neurologic exam, and brain magnetic resonance imaging (MRI) with contrast were obtained after each cycle. Toxicity assessments were obtained after each cycle. Toxicity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0.

SCHEDULE OF EVENTS - PROTOCOL ACTIVITIES

<14 Days Prior to Initial Study Treatment:

* Neurological/Oncological History
* Neurological Examination
* Height/Weight/Body Surface Area
* Performance Status
* Quality of Life (QOL) FACT-L
* Laboratory Studies; complete blood count (CBC), Differential, Platelets, prothrombin time/partial thromboplastin time (PT/PTT), international normalized ratio (INR), Serum Creatinine, blood urea nitrogen (BUN), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactate dehydrogenase (LDH), Total Bilirubin, alkaline phosphatase (AlkPHs), Pregnancy Test, electrocardiogram (EKG)
* Cranial MRI or CT with and without contrast
* Multiple uptake gated acquisition (MUGA) Scan

Day 1, At the Beginning of Each Treatment Cycle:

* Adverse Event Assessment
* Laboratory Studies; CBC, Differential, Platelets

Every Cycle, Days 42-45 (within 3 days of next scheduled Sutent treatment):

* Neurological/Oncological History
* Neurological Examination
* Height/Weight/Body Surface Area
* Performance Status
* QOL FACT-L
* Laboratory Studies; Serum Creatinine, BUN, ALT, AST, LDH, Total Bilirubin, AlkPHs
* Cranial MRI or CT with and without contrast
* Survival

At Off Study:

* Performance Status
* Cranial MRI or CT with and without contrast
* Survival

ELIGIBILITY:
Inclusion Criteria:

* Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade ≤1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤3 x local laboratory upper limit of normal (ULN), or AST and ALT ≤3 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin ≤1.5 x ULN
  * Absolute neutrophil count (ANC) ≥1500/µL
  * Platelets ≥100,000/µL
  * Hemoglobin ≥9.0 g/dL
  * Serum calcium ≤12.0 mg/dL
  * Serum creatinine ≤1.5 x ULN
* Patients must have histologically or neuroradiographically recurrent anaplastic astrocytoma (AA) or glioblastoma (GBM). Must have had prior pathologic confirmation of primary tumor histology.
* Must be ≥ 18 years old.
* Must have a Karnofsky performance status (KPS) ≥ 60%
* Measurable disease per MacDonald criteria required using contrast enhanced cranial MRI.
* Life expectancy ≥ 12 weeks.
* Must sign and date an Institutional Review Board (IRB) approved informed consent stating that he or she is aware of the neoplastic nature of the disease. Must willingly provide written consent after being informed of procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and accessible for follow-up.
* Have undergone surgery documenting tumor histology though repeat surgery at time of tumor recurrence is not mandatory.
* Have received prior external beam radiotherapy.
* Patients may have received one or two prior salvage chemotherapy and may have received adjuvant chemotherapy following initial surgery.
* May not have received prior stereotactic radiotherapy.
* May have been treated with Gliadel at initial surgery only.

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks of starting study treatment.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting study treatment.
* History of or known spinal cord compression or carcinomatous meningitis, or evidence of leptomeningeal disease on screening CT or MRI scan.
* Any of the following within 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
* Prolonged QTc interval on baseline EKG.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in normal range with medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Concomitant use of ketoconazole and other agents known to inhibit Cytochrome P450 3A4 (CYP3A4).
* Concomitant use of theophylline and phenobarbital and/or other agents metabolized by the cytochrome P450 system.
* Ongoing treatment with therapeutic doses of Coumadin (low dose up to 2 mg po daily for thrombo-prophylaxis is allowed).
* Pregnancy or breastfeeding. Female subjects must be surgically sterile, postmenopausal, or must agree to use effective contraception during the period of therapy. Female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with interpretation of study results, and in the judgment of investigator would make patient inappropriate for entry into this study.
* Patients having been treated with 3 or more salvage regimens.
* Patients with a second active malignancy or diagnosis of other cancer within 3 years of enrollment, except for surgically cured basal cell carcinoma, or in situ carcinoma of the cervix.
* Mentally incapacitated patients or psychiatric illness that would prevent them from giving informed consent.
* Poorly controlled diabetes, hepatitis infection, uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, and myocardial infarction within previous 6 months, or serious uncontrolled cardiac arrhythmia.
* Known to be HIV positive or to have an AIDS-related illness.
* Patients with an active infection that is not adequately controlled with antibiotics.
* Patients with other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Known sensitivity to any of the products to be administered during treatment.
* Currently enrolled in another clinical trial or patients who have participated in a trial of an investigational device or drug within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients must have had pathologically or neuroradiographically recurrent AA or GB and prior pathologic confirmation of primary tumor histology. Patients with prior low-grade glioma were eligible if histological transformation to malignant astrocytic gliomas (MAG) was confirmed before enrollment.
Pre-assignment Details: Study patients were stratified by tumor histology (AAor GB).
Groups:
- Sutent Treatment: Sutent was administered daily for 4 weeks at a dose of 50 mg followed by a 2 week study drug free break.
  Sunitinib Malate : Initially, patients were started on sunitinib at a dose of 50 mg daily. If 50 mg daily resulted in unacceptable toxicity, 2 dose modifications were allowed (to 37.5 and to 25 mg daily, if necessary). Study patients who could not tolerate 25 mg daily of sunitinib were taken off study.
Period: Overall Study
Arm/Group | Sutent Treatment
Started | 30
Completed | 25
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sutent Treatment
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Age Continuous [Median (Full Range); unit: years] | 52 [30.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months Utilizing McDonald Criteria for Response, Progression and Relapse
Description: Complete Response: Disappearance of all lesions, disease signs and symptoms related to the tumor. Partial Response (PR): When compared with pretreatment measurements, a reduction of 50% decrease in the sum of the longest diameters of all target enhancing lesions, taking as reference the baseline sum of the longest diameter. Stable Disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameter since treatment started. Objective Progression or Relapse: Relative to pretreatment measurements, an increase in the sum of the diameters of any measured enhancing lesion by at least 25% increase in the sum of the longest diameters since the treatment started or the appearance of new enhancing lesions.
Time Frame: 6 Months
Population: All participants
Measure: Number; unit: Participants
Groups:
- AA Cohort Patients: Recurrent glioblastoma (GB) patients
- GB Cohort Patients: Anaplastic astrocytoma (AA)patients
Arm/Group | Sutent Treatment | AA Cohort Patients | GB Cohort Patients
Number analyzed (Participants) | 30 | 14 | 16
Participants | 4 | 2 | 2

2. Secondary Outcome: Best Overall Response
Description: To estimate best response rates (proportion of patients who ever had a radiographic response equal to or better than stable disease during course assessment).
Time Frame: 12 Months
Population: All participants
Measure: Number; unit: Participants
Arm/Group | Sutent Treatment | AA Cohort Patients | GB Cohort Patients
Number analyzed (Participants) | 30 | 14 | 16
Participants | 13 | 8 | 5

3. Secondary Outcome: Number of Participants With Related Grade 3 and Greater Adverse Events
Description: To evaluate toxicities associated with sunitinib treatment (grade 3 and greater toxicities).
Time Frame: 12 Months
Population: All participants
Measure: Number; unit: Participants
Arm/Group | Sutent Treatment | AA Cohort Patients | GB Cohort Patients
Number analyzed (Participants) | 30 | 14 | 16
Participants | 11 | 6 | 5

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Description: Toxicity assessments were obtained after each cycle. Toxicity was graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Response evaluations were performed using modified Macdonald criteria. Serious Adverse Events: =/> Grade 3 toxicities associated with sunitinib.
Arm/Group | Sutent Treatment | AA Cohort Patients | GB Cohort Patients
Serious Adverse Events (participants affected / at risk) | 11/30 | 6/14 | 5/16
Other Adverse Events (participants affected / at risk) | 28/30 | 14/14 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sutent Treatment (N=30) | AA Cohort Patients (N=14) | GB Cohort Patients (N=16)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Platelets (Blood and lymphatic system disorders) | 4 | 2 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 | 1 | 2
Death not associated with CTCAE term - disease progression NOS (General disorders) | 1 | 1 | 0
Dermatology/skin-other (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Hemorrhage/bleeding-other (General disorders) | 1 | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 0 | 1
Mucositis/stomatitis (functional/symptomatic) - anus (Gastrointestinal disorders) | 1 | 0 | 1
ALT, SGPT (Metabolism and nutrition disorders) | 1 | 0 | 1
AST, SGOT (Metabolism and nutrition disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sutent Treatment (N=30) | AA Cohort Patients (N=14) | GB Cohort Patients (N=16)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21 (27) | 11 (12) | 10 (15)
Dermatology/Skin - other (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (5) | 3 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8) | 2 (2) | 5 (6)
Ataxia (incoordination) (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Confusion (General disorders) | 4 (5) | 3 (3) | 1 (2)
Mood alteration - Depression (General disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy: cranial - CN IV Downward, inward movement of eye (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Pain - Back (General disorders) | 3 (3) | 2 (2) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 1 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Weight loss (General disorders) | 4 (4) | 2 (2) | 0 (0)
Lymphatics - other (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1)
Gastrointestinal - other (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (8) | 5 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Cognitive disturbance (General disorders) | 3 (3) | 2 (2) | 1 (2)
Neuropathy: cranial - CN II Vision (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 11 (13) | 5 (6) | 6 (7)
Neuropathy: sensory (Nervous system disorders) | 8 (10) | 5 (6) | 3 (4)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 5 (5) | 2 (2) | 3 (3)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 (7) | 3 (5) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7 (13) | 4 (6) | 3 (7)
Platelets (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (16) | 7 (8) | 8 (8)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity - lower (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity - upper (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain - Head/headache (Nervous system disorders) | 8 (10) | 2 (3) | 6 (7)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4) | 2 (2)
Insomnia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Muscoleoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 (6) | 2 (2) | 3 (4)
Seizure (Nervous system disorders) | 3 (4) | 2 (3) | 1 (1)
Pain - Abdomen NOS (General disorders) | 2 (2) | 0 (0) | 2 (2)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Pain - Other (General disorders) | 3 (3) | 1 (1) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 1 (3)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Vision - Blurred vision (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Pain - Stomach (General disorders) | 2 (2) | 0 (0) | 2 (2)
Perforation, GI - Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Mucosa (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sweating (diaphoresis) (General disorders) | 4 (5) | 2 (2) | 2 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy: cranial - CN VII Motor-face; Sensory-taste (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Hearing: patients without baseline audiogram and not enrolled n a monitoring program (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (4) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (5) | 1 (3) | 2 (2)
Hypertension (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy: cranial - CN I Smell (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy: cranial - CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pain - Extremity-limb (General disorders) | 2 (3) | 1 (1) | 1 (2)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Allergy/Immunology - Other (Immune system disorders) | 3 (3) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Infection with unknown ANC - Lung pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) - Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection with unknown ANC - Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain - Chest wall (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain - Eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Mood alteration - Agitation (General disorders) | 5 (5) | 3 (3) | 2 (2)
Hemorrhage/Bleeding - Other (General disorders) | 1 (1) | 0 (0) | 1 (1)
Neurology - Other (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
No definitive conclusions can be made regarding outcome differences between bevacizumab vs. bevacizumab-naive study patients, due to not enough patients who received bevacizumab prior to study enrollment (2 AA, 3 GB).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes